CLINICAL TRIAL: NCT06104813
Title: Evaluation of Deaf Men's Knowledge About Sexual Health, in Nancy's CHRU
Brief Title: Evaluation of Deaf Men's Knowledge About Sexual Health
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, BOUILLEVAUX Isabelle, Doctor Bouillevaux Isabelle, Central Hospital, Nancy, France
Other Study IDs: 2022PI188-398
Record Dates: First submitted 2023-10-24; First posted 2023-10-27 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Deafness; Sexual Satisfaction; Sexually Transmitted Diseases; Sexual Violence; Educational Problems
Keywords: Deafness; Sexual Health; Sexually Transmitted Diseases; Sexual Violence; Sexual Health Awareness
MeSH Terms: conditions — Deafness; Orgasm; Sexually Transmitted Diseases | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- URASSM volunteer deaf men: Volunteer deaf men recruited at Nancy's URASSM Deaf Care Unit (Unité régionale d'accueil et de soins des sourds et malentendants), for individual interviews.
  Interventions: Other: Interviews

INTERVENTIONS:
Other: Interviews — Interview with volunteer, to ask them a series of open questions about sexual health in the deaf male population.

SUMMARY:
Evaluation of Deaf men's knowledge about sexual health in Nancy, France. The study consists of interviews with voluntary deaf men from Nancy, France, in order to assess their knowledge about sexual health, and determine if there is a lack of sexual health awareness.

If there is indeed a lack of information about sexual health, the study aims at finding ways of improving the situation, and see how the deaf men would like to have this information delivered to them.

DETAILED DESCRIPTION:
Evaluation of Deaf men's knowledge about sexual health in Nancy, France. The study consists of interviews with voluntary deaf men from Nancy, France. The goal is to assess their knowledge about sexual health, and determine if there is a lack of sexual health awareness.

If there is indeed a lack of information about sexual health, the study aims at finding ways of improving the situation, and see how the deaf men would like to have sexual health information delivered to them.

Patients from Nancy's Regional Deaf Healthcare Service (URASSM) will be contacted and volunteers adult deaf men, using sign language as their main langage, will be recruited into the study.

The interviews will consist of a series of open questions aiming to evaluate the volunteers knowledge about sexual health, and evaluate their expectations about how sexual health care for deaf men should be dealt with.

A professional french sign language translator will be present during the interviews, and all the questions and answers will be delivered using french sign language.

ELIGIBILITY:
Inclusion Criteria:

* Deaf
* Over 18
* Using french sign language
* Whithout curatorship or tutelage

Exclusion Criteria:

* Female
* Under 18
* Non deaf

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Volunteer deaf men over 18 whitout curatorship or tutelage, using french signe language as their main language.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2023-09-11 (Actual); Primary Completion 2023-10-23 (Actual); Study Completion 2023-10-23 (Actual)

PRIMARY OUTCOMES:
Deaf volunteer's sexual health knowledge questionnaire | 1 day Interview
  Deaf volunteer's sexual health knowledge about sexual violence, STDS, contraceptives

SECONDARY OUTCOMES:
Deaf volunteer's expectation about sexual health care questionnaire | 1 day Interview
  Deaf volunteer's expectation about sexual health care, especially how they would like to get information delivered to them, and how a medical consultation dealing with sexual health should be performed.

CONTACTS AND LOCATIONS:
Locations (1):
- Central Hospital, Nancy, Grand Est, France

IPD SHARING:
Plan to Share IPD: No